CLINICAL TRIAL: NCT01496170
Title: A Study to Assess the Safety, Tolerability, and Pharmacodynamics of MK-8931/SCH 900931 in Patients With Alzheimer's Disease [Phase 1b; Protocol No. 010-00 (Also Known as P07820)]
Brief Title: A Study of the Safety, Tolerability, and Pharmacodynamics of MK-8931 in Participants With Alzheimer's Disease (MK-8931-010 AM1 [P07820 AM1])
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P07820; MK-8931-010 (Other: Schering-Plough)
Record Dates: First submitted 2011-12-06; First posted 2011-12-21 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — verubecestat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A: MK-8931 12 mg (Experimental): Participants receiving 12 mg MK-8931 for 7 days
  Interventions: Drug: MK-8931
- Treatment B: MK-8931 40 mg (Experimental): Participants receiving MK-8931 40 mg for 7 days
  Interventions: Drug: MK-8931
- Treatment C: Placebo matching MK-8931 12 mg or 40 mg (Placebo Comparator): Participants receiving placebo matching MK-8931 12 mg or 40 mg for 7 days
  Interventions: Drug: Placebo
- Treatment D: MK-8931 60 mg (Experimental): Participant receiving MK-8931 60 mg for 7 days
  Interventions: Drug: MK-8931
- Treatment E: Placebo matching MK-8931 60 mg (Placebo Comparator): Participants receiving placebo matching MK-8931 60 mg for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8931 — MK-8931, capsules, at a dose of 12 or 40 mg, orally, once per day for 7 days
  Other Names: SCH 900931
  Arms: Treatment A: MK-8931 12 mg; Treatment B: MK-8931 40 mg; Treatment D: MK-8931 60 mg
Drug: Placebo — Placebo capsules, orally, once per day for 7 days
  Arms: Treatment C: Placebo matching MK-8931 12 mg or 40 mg; Treatment E: Placebo matching MK-8931 60 mg

SUMMARY:
This study will assess the safety and pharmacodynamics of three different doses of MK-8931, a ß-secretase inhibitor, in participants with mild to moderate Alzheimer's Disease (AD).

ELIGIBILITY:
Inclusion criteria:

* Body Mass Index (BMI) between 18 and 35
* Mild to moderate Alzheimer's Disease (AD)
* Clear history of cognitive and functional decline over at least one year that is either documented in medical records, or documented by history from an informant who knows the subject well
* Magnetic Resonance Image (MRI) scan consistent with a diagnosis of AD
* Ability to read at a 6th grade level and history of academic achievement and/or employment sufficient to exclude mental retardation
* If applicable, on a stable dose of an acetylcholinesterase inhibitor and/or memantine for at least the last 3 months before Screening, and willing to remain on the same dose for the duration of the trial
* Reliable trial partner/caregiver
* Willing to provide a blood sample for Apolipoprotein E (APOE) genotyping
* In general good health (other than AD)
* Participant capable of conceiving and/or participant with partner capable of conceiving willing to use a medically acceptable form of contraception during the trial and for 3 months after stopping the medication

Exclusion criteria:

* History (within 2 years of the prestudy visit) or current evidence of any neurological or neurodegenerative disorder other than AD that is associated with transient or sustained alterations in cognition
* Clinically significant abnormalities in serum vitamin B12, folate, thyroid stimulating hormone (TSH) or thyroxin 4 (T4). Vitamin B12 or thyroid replacement therapy must with stable dose for at least 2 months prior to screening visit
* One or more pre-existing risk factors for Torsades de Pointes: New York Heart Association (NYHA) Functional Classification II through IV heart failure; Familial Long QT Syndrome; or Uncorrected hypokalemia
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug
* History of spinal cord compression or any other current abnormalities in the lumbar region (skin infection, developmental abnormalities in lower spine, etc.)
* History of any infectious disease within 4 weeks prior to drug administration
* Human immunodeficiency virus (HIV) positive
* History of hepatitis or liver disease within 6 months of screening
* History of psychiatric or personality disorders
* Evidence of suicidality or is at risk for self-harm or harm to others
* History of seizures or epilepsy or anticonvulsant use within the last 5 years before Screening
* History of alcohol or drug abuse in the past 2 years
* Donation of blood in the past 60 days
* Previously received the study drug
* Currently participating in another clinical study or have participated in a clinical study (e.g., laboratory or clinical evaluation) within 30 days of baseline
* Member of the study staff or family members of the study staff
* Demonstrated allergic reactions (e.g., food, drug, atopic reactions or asthmatic episodes)
* History of malignancy occurring within the 5 years immediately before Screening, except for a subject who has been adequately treated for basal cell or squamous cell skin cancer, in situ cervical cancer, localized prostate carcinoma; or has undergone potentially curative therapy with no evidence of recurrence for ≥1 year post-therapy, and deemed at low risk for recurrence by her/his treating physician

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Mean population Inhibitory Concentration for 50% Effect (IC50) in cerebral spinal fluid (CSF) ß-amyloid peptide 40 (Aß40) | Hour 0 (predose) to 36 hours post-dose on Day 7

SECONDARY OUTCOMES:
Change in CSF Aß40 concentration determined by time-weighted average from 0 to 24 hours (TWA0-24) | Baseline, and assessment over 24 hours post Day 7 dose
Change in CSF soluble amyloid precursor protein ß (sAPPß ) concentration determined by TWA0-24 | Baseline, and assessment over 24 hours post Day 7 dose

REFERENCES:
- [Derived] Kennedy ME, Stamford AW, Chen X, Cox K, Cumming JN, Dockendorf MF, Egan M, Ereshefsky L, Hodgson RA, Hyde LA, Jhee S, Kleijn HJ, Kuvelkar R, Li W, Mattson BA, Mei H, Palcza J, Scott JD, Tanen M, Troyer MD, Tseng JL, Stone JA, Parker EM, Forman MS. The BACE1 inhibitor verubecestat (MK-8931) reduces CNS beta-amyloid in animal models and in Alzheimer's disease patients. Sci Transl Med. 2016 Nov 2;8(363):363ra150. doi: 10.1126/scitranslmed.aad9704. PMID 27807285